CLINICAL TRIAL: NCT06806904
Title: The Role of Ultrasonography in Labor in Predicting the Outcomes of Childbirth
Acronym: EcoSP_21
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EcoSP_21
Record Dates: First submitted 2024-12-30; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Ultrasound in Labor
Keywords: labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ultrasound in the delivery room represents a useful diagnostic tool and is used for the assessment of fetal presentation, fetal malpresentation/malposition, and prior to any operative delivery. Transperineal ultrasonography, performed by placing the ultrasound probe covered by a sterile glove at the level of the labia majora, has proven useful in providing information on the progression of the presented fetal part in the birth canal and in predicting birth outcomes. Many studies have shown a correlation between the above ultrasound indices and birth outcomes. These ultrasound indices are therefore used in clinical practice to assess the progression of the presented fetal part in the birth canal and the presence of fetal malpresentation/malposition. Despite this, to date, few studies have evaluated the correlation between dynamic changes in these ultrasound parameters between rest and maximal maternal pushing during the second stage of labor and birth outcomes.

Knowing before delivery which parameters are suggestive of possible dystocia would allow the clinician to adopt therapeutic strategies aimed at resolving them and thus increase the rate of spontaneous vaginal deliveries.

The investigators want to evaluate the role of an ultrasound parameter obtained by transabdominal ultrasound in the second stage of labor, the occiput-column angle, in predicting spontaneous delivery vaginally in fetuses with transverse occiput

DETAILED DESCRIPTION:
Participants will be recruited at the time of admission or in the delivery room. Routine clinical practice involves transabdominal ultrasound, performed in the lithotomy position, placing the probe transversely and longitudinally at the abdominal level for evaluation of the fetal situation and presentation.

In addition to normal ultrasound, the position of the fetal occiput will also be assessed in women who agree to participate in the study, and in fetuses with a transverse occiput, the occipitecolumn angle will be measured. All study participants will then undergo transperineal ultrasound, performed by placing the probe, covered by a sterile glove, at the level of the labia majora, first longitudinally and then transversely. In this way, a series of ultrasound landmarks will be visualized: pubic symphysis, bladder, urethra, vagina, rectum, pubo-rectal muscle, and fetal head.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >= 18 years
* Single pregnancy at term (37-42 gestational weeks)
* Fetus in cephalic presentation and in expulsive period (complete cervical dilatation and premature sensation)
* Acquisition of informed consent form

Exclusion Criteria:

* Placenta previa
* Uterine malformations
* Previous uterine surgery
* Cardiotocographic tracing (CTG) abnormalities
* Any contraindication to vaginal delivery

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: It is planned to enroll patients afferent to the Department of Obstetrics and Prenatal Age Medicine, Sant'Orsola-Malpighi Polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of Angle of Progression (AoP) | At the time of delivery: at rest and during maternal pushing
  Angle of progression (AoP): the angle between the longitudinal axis of the pubic symphysis and a straight line starting from the lower edge of the symphysis and passing tangentially to the most distal part of the fetal head
Measurement of Anteroposterior Pelvic Hiatus Diameter (APD) | At the time of delivery: at rest and during maternal pushing
  Anteroposterior pelvic hiatus diameter (APD): distance between the posteroinferior margin of the pubic symphysis and the anterior margin of the pubo-rectal muscle
Measurement of Head-Sympanic Distance (HSD) | At the time of delivery: at rest and during maternal pushing
  Head-symphysis distance (HSD): distance between the lower edge of the pubic symphysis and the nearest point of the fetal scalp along the infrapubic line
Measurement of Head-Perineum Distance (HPD) | At the time of delivery: at rest and during maternal pushing
  Head-Perineum Distance (HPD): distance between the perineum and the nearest point of the fetal scalp

CONTACTS AND LOCATIONS:
Overall Officials: Aly Mohamed Alaaeldin Kamaleldin Aly Youssef, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy